CLINICAL TRIAL: NCT05631184
Title: Self-administered Acupressure for Depression: A Randomized Controlled Trial
Brief Title: Self-administered Acupressure for Depression
Acronym: SAAFD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SelfAcupDep; 19200171 (Other Grant/Funding Number: Health and Medical Research Fund)
Record Dates: First submitted 2022-11-14; First posted 2022-11-30 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Depressive Symptoms; Depressive Disorder; Depression
Keywords: Depression; Acupressure; Randomized Controlled Trial
MeSH Terms: conditions — Depression; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment involves two groups of participants. In this study, one group will receive self-administered acupressure, and the other group will receive the mental health education. So during the trial, participants in one group receive self-administered acupressure "in parallel" to participants in the other group, who receive the mental health education.
Who Masked: Outcomes Assessor
Masking Description: The researchers who perform the assessment and analysis will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-administered acupressure group (Experimental): The participants in the self-administered acupressure group will attend an acupressure training course (2 sessions, 2 h each) to learn self-administered acupressure from an acupuncturist in a classroom at the School Nursing, the Hong Kong Polytechnic University. Each class will be conducted in a small group of 4 to 7 participants to enhance interaction and ensure the quality of teaching. Participants will then practice two times a day for 8 weeks.
  Interventions: Behavioral: Self-administered acupressure group
- Mental health education group (Active Comparator): The participants in the comparison group will receive mental health education group from a registered nurse with the same frequency as those in the treatment group (2 sessions, 2 h each) in a classroom at the School Nursing, the Hong Kong Polytechnic University, and will be reminded to follow the mental health practice daily for 8 weeks.
  Interventions: Behavioral: Mental health education group

INTERVENTIONS:
Behavioral: Self-administered acupressure group — Self-administered acupressure treatment group was developed on the basis of previous systematic reviews and clinical studies of acupuncture and acupressure for depression. It has robust theoretical basis of TCM. The acupoints selected are commonly used for depression according to a recent systematic review and recommended by other clinical practice guidelines.
  Arms: Self-administered acupressure group
Behavioral: Mental health education group — Mental health education training group was developed based on the materials regarding depression and mental health from the Centre of Health Protection, Department of Health, the Government of Hong Kong SAR and reviewed by a clinical psychologist.
  Arms: Mental health education group

SUMMARY:
The goal of this clinical trial is to examine the effects of self-administered acupressure intervention for alleviating depressive symptoms among people with depression. It is hypothesized that the self-administered acupressure group would have a great improvement in depressive symptoms as measured by the Patient Health Questionnaire compared with the mental health education group across the 12-week intervention period.

The main questions it aims to answer are:

* Is the self-administered acupressure intervention more effective for alleviating depression and other related outcomes compared to the mental health education group among depressed individuals?
* Is the self-administered acupressure intervention acceptable and feasible for depressed individuals to alleviate depression? Participants will be randomized into self-administered acupressure group or mental health education group based on the group allocation with a 1:1 ratio. Participants will attend two weekly 120-min self-administered acupressure training or mental health education, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged 18 to 65
2. Can communicate in Cantonese and comprehend written Chinese
3. Have moderate or above-level depression as measured by the PHQ-9 with a score of 10 or above
4. Willing to give informed consent and comply with the trial protocol.

Exclusion Criteria:

1. Have the PHQ score of 20 or above (referral information to community psychological services will be provided)
2. New onset or change of antidepressant medication or dosage in the last 3 months
3. Previous or current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder as screened using the Chinese version of the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders.
4. Have cognitive impairment diagnosed by the Hong Kong Montreal Cognitive Assessment with a score < 22
5. Skin lesions or infections at the treatment sites
6. Significant suicidal risk as rated by the Hamilton Depression Rating Scale item on suicide (score ≥3)
7. Pregnant or childbearing potential but not using adequate contraception
8. With any major medical condition that causes depression based on the judgement of a psychiatrist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ) | It will be measured at baseline
  The PHQ-9, a self-rated questionnaire to assess depressive symptoms over the last 2 weeks on a scale of 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 27.
Patient Health Questionnaire (PHQ) | It will be measured at week 4 from baseline
  The PHQ-9, a self-rated questionnaire to assess depressive symptoms over the last 2 weeks on a scale of 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 27.
Patient Health Questionnaire (PHQ) | It will be measured at week 8 from baseline
  The PHQ-9, a self-rated questionnaire to assess depressive symptoms over the last 2 weeks on a scale of 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 27.
Patient Health Questionnaire (PHQ) | It will be measured at week 12 from baseline
  The PHQ-9, a self-rated questionnaire to assess depressive symptoms over the last 2 weeks on a scale of 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 27.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | It will be measured at baseline
  The HDRS is used to assess the severity of depressive symptoms based on the 17-item scale. Eight items are scored on a 5-point scale, ranging from 0 to 4 and nine items are scored from 0 to 2. The total score varies from 0 (the minimum value) to 52 (the maximum value), with a higher total score indicating more severe depression.
Hamilton Depression Rating Scale (HDRS) | It will be measured at week 4 from baseline
  The HDRS is used to assess the severity of depressive symptoms based on the 17-item scale. Eight items are scored on a 5-point scale, ranging from 0 to 4 and nine items are scored from 0 to 2. The total score varies from 0 (the minimum value) to 52 (the maximum value), with a higher total score indicating more severe depression.
Hamilton Depression Rating Scale (HDRS) | It will be measured at week 8 from baseline
  The HDRS is used to assess the severity of depressive symptoms based on the 17-item scale. Eight items are scored on a 5-point scale, ranging from 0 to 4 and nine items are scored from 0 to 2. The total score varies from 0 (the minimum value) to 52 (the maximum value), with a higher total score indicating more severe depression.
Hamilton Depression Rating Scale (HDRS) | It will be measured at week 12 from baseline
  The HDRS is used to assess the severity of depressive symptoms based on the 17-item scale. Eight items are scored on a 5-point scale, ranging from 0 to 4 and nine items are scored from 0 to 2. The total score varies from 0 (the minimum value) to 52 (the maximum value), with a higher total score indicating more severe depression.
The Depression Anxiety Stress Scales (DASS-21) - Stress | It will be measured at baseline
  The DASS-21 Stress subscale will be used to measure the emotional states of stress using a 4-point scale ranging from 0 (never) to 3 (almost always).
The Depression Anxiety Stress Scales (DASS-21) - Stress | It will be measured at week 4 from baseline
  The DASS-21 Stress subscale will be used to measure the emotional states of stress using a 4-point scale ranging from 0 (never) to 3 (almost always).
The Depression Anxiety Stress Scales (DASS-21) - Stress | It will be measured at week 8 from baseline
  The DASS-21 Stress subscale will be used to measure the emotional states of stress using a 4-point scale ranging from 0 (never) to 3 (almost always).
The Depression Anxiety Stress Scales (DASS-21) - Stress | It will be measured at week 12 from baseline
  The DASS-21 Stress subscale will be used to measure the emotional states of stress using a 4-point scale ranging from 0 (never) to 3 (almost always).
The Depression Anxiety Stress Scales (DASS-21) - Anxiety | It will be measured at baseline
  The DASS-21 Anxiety subscale will be used to measure the emotional states of anxiety using a 4-point scale ranging from 0 (never) to 3 (almost always).
The Depression Anxiety Stress Scales (DASS-21) - Anxiety | It will be measured at week 4 from baseline
  The DASS-21 Anxiety subscale will be used to measure the emotional states of anxiety using a 4-point scale ranging from 0 (never) to 3 (almost always).
The Depression Anxiety Stress Scales (DASS-21) - Anxiety | It will be measured at week 8 from baseline
  The DASS-21 Anxiety subscale will be used to measure the emotional states of anxiety using a 4-point scale ranging from 0 (never) to 3 (almost always).
The Depression Anxiety Stress Scales (DASS-21) - Anxiety | It will be measured at week 12 from baseline
  The DASS-21 Anxiety subscale will be used to measure the emotional states of anxiety using a 4-point scale ranging from 0 (never) to 3 (almost always).
The Insomnia Severity Index (ISI) | It will be measured at baseline
  The ISI is a seven-item self-rating scale to assess the severity of insomnia, distress, and functional impairment associated with insomnia on a 5-point Likert scale.
The Insomnia Severity Index (ISI) | It will be measured at week 4 from baseline
  The ISI is a seven-item self-rating scale to assess the severity of insomnia, distress, and functional impairment associated with insomnia on a 5-point Likert scale.
The Insomnia Severity Index (ISI) | It will be measured at week 8 from baseline
  The ISI is a seven-item self-rating scale to assess the severity of insomnia, distress, and functional impairment associated with insomnia on a 5-point Likert scale.
The Insomnia Severity Index (ISI) | It will be measured at week 12 from baseline
  The ISI is a seven-item self-rating scale to assess the severity of insomnia, distress, and functional impairment associated with insomnia on a 5-point Likert scale.
The Short-Form (six-dimension) Health Survey (SF-6D) | It will be measured at baseline
  The SF-6D covers six domains using a scale of 1 to 6 to evaluate participants' general health and quality of life.
The Short-Form (six-dimension) Health Survey (SF-6D) | It will be measured at week 4 from baseline
  The SF-6D covers six domains using a scale of 1 to 6 to evaluate participants' general health and quality of life.
The Short-Form (six-dimension) Health Survey (SF-6D) | It will be measured at week 8 from baseline
  The SF-6D covers six domains using a scale of 1 to 6 to evaluate participants' general health and quality of life.
The Short-Form (six-dimension) Health Survey (SF-6D) | It will be measured at week 12 from baseline
  The SF-6D covers six domains using a scale of 1 to 6 to evaluate participants' general health and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Wing Fai Yeung, PhD, Principal Investigator — the School of Nursing, the Hong Kong Polytechnic University
Locations (1):
- School of Nursing, the Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available when the study has been published. The individual participant data will be available upon request.
Supporting Information: Study Protocol, SAP
Time Frame: No time restriction for the data availability.
Access Criteria: The individual participant data will be available upon request.

REFERENCES:
- [Background] Zhang Z, Li S, Meng H, Wang Y, Zhang Y, Wu M, Chen Y, Rong P, Wang Y. Efficacy and safety of acupuncture in the treatment of depression: A systematic review of clinical research. Anat Rec (Hoboken). 2021 Nov;304(11):2436-2453. doi: 10.1002/ar.24783. Epub 2021 Oct 8. PMID 34623754
- [Background] Fernandez-Chinguel JE, Goicochea-Lugo S, Villarreal-Zegarra D, Taype-Rondan A, Zafra-Tanaka JH. Acupuncture for major depressive disorder: A review of the recommendations stated at clinical practice guidelines. Complement Ther Med. 2020 Mar;49:102321. doi: 10.1016/j.ctim.2020.102321. Epub 2020 Jan 24. PMID 32147048
- [Background] Cheung DST, Tiwari A, Yeung WF, Yu DSF, So MKP, Chau PH, Wang XM, Lum TYS, Yuk Fung HYK, Ng BYM, Zhang ZJ, Lao L. Self-Administered Acupressure for Caregivers of Older Family Members: A Randomized Controlled Trial. J Am Geriatr Soc. 2020 Jun;68(6):1193-1201. doi: 10.1111/jgs.16357. Epub 2020 Feb 25. PMID 32096884
- [Background] Kroenke K. Enhancing the clinical utility of depression screening. CMAJ. 2012 Feb 21;184(3):281-2. doi: 10.1503/cmaj.112004. Epub 2012 Jan 9. No abstract available. PMID 22231681